CLINICAL TRIAL: NCT00707642
Title: Phase 1, Open-Label, Safety Study of HBV-002 (West Nile Recombinant Subunit Vaccine) in Healthy Adults
Brief Title: Safety Study of HBV-002 West Nile Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hawaii Biotech, Inc. (Industry)
Responsible Party: Beth-Ann Coller, Ph.D., Hawaii Biotech
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HBV-002-C-101
Record Dates: First submitted 2008-06-29; First posted 2008-07-01 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: West Nile Virus Disease
Keywords: West Nile Virus; West Nile Vaccine; West Nile virus disease; Hawaii Biotech

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Low Dose WN-80E API (5 µg) + Alhydrogel (3.5 mg)
  Interventions: Biological: WN-80E
- 2 (Experimental): Medium Dose WN-80E API (15 µg) + Alhydrogel (3.5 mg)
  Interventions: Biological: WN-80E
- 3 (Experimental): High Dose WN-80E API (50 µg) + Alhydrogel (3.5 mg)
  Interventions: Biological: WN-80E
- 4 (Experimental): High Dose WN-80E API (50 µg), no adjuvant
  Interventions: Biological: WN-80E

INTERVENTIONS:
Biological: WN-80E — Three injections of the study vaccine [Low Dose of WN-80E API (5 µg) + Alhydrogel (3.5 mg)] given one month apart
  Other Names: HBV-002 vaccine
  Arms: 1
Biological: WN-80E — Three injections of the study vaccine [Medium Dose WN-80E API (15 µg) + Alhydrogel (3.5 mg)] given one month apart
  Other Names: HBV-002 vaccine
  Arms: 2
Biological: WN-80E — Three injections of the study vaccine [High Dose WN-80E API (50 µg) + Alhydrogel (3.5 mg)] given one month apart
  Other Names: HBV-002 vaccine
  Arms: 3
Biological: WN-80E — Three injections of the study vaccine [High Dose WN-80E API (50 µg)] given one month apart
  Other Names: HBV-002 vaccine
  Arms: 4

SUMMARY:
The purpose of this Phase 1 trial is to evaluate the clinical safety of HBV-002 vaccine in healthy adults.

DETAILED DESCRIPTION:
West Nile virus is an emerging infectious disease in the U.S. and worldwide and has been identified by the CDC as a significant public health risk. Since the introduction of West Nile virus into the U.S. in 1999, annual outbreaks have caused severe and fatal encephalitis in humans and equines and death in a variety of species of feral birds throughout the U.S. and parts of Canada. In addition, more recent findings show evidence of West Nile virus human and equine infection in several countries of tropical America. The virus has now been found in bird populations in all 48 states of the continental U.S, and human cases of West Nile disease have been documented in 45 states and the District of Columbia. To date, there is no approved commercial vaccine available for prevention of West Nile virus disease in humans.

ELIGIBILITY:
Inclusion Criteria:

* Satisfactory medical assessment with no clinically significant and relevant abnormalities (medical history, physical examination, vital signs, ECG, clinical laboratory evaluation [hematology, biochemistry, urinalysis])
* Body weight must not be more than 10% below of 20% above the ideal weight for height and frame size according to the 1999 Metropolitan Life table

Exclusion Criteria:

* Current active infection process including URI or influenza
* Positive serum test for HIV, Hepatitis B surface antigens and/or Hepatitis C antibodies
* History of infection with, or serologic evidence in screening test, of prior flavivirus infection (to include viruses: West Nile, 4 dengue serotypes, yellow fever (YF), and Japanese encephalitis (JE)
* Subject has resided in flavivirus (West Nile, 4 dengue serotypes, YF, and JE) endemic areas or has a history of receipt of Yellow Fever or Japanese encephalitis virus vaccines
* History of alcohol or other substance abuse within 1 year of screening
* Use of corticosteroids or immunosuppressive drugs within 30 days of screening (Use of topical or nasal corticosteroids are not excluded.)
* Any confirmed or suspected immunosuppressive or immunodeficient condition
* Administration of immunoglobulins within three months of the first vaccination or planned during the study period
* Receipt of any vaccines or investigational or non-registered product other than HBV-002 within 30 days prior to screening or planned receipt throughout the study.
* Receipt of another study vaccines within 30 days prior to screening
* Receipt of blood products within 6 months of screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of the study HBV-002 formulations in healthy adult subjects | 38 weeks

SECONDARY OUTCOMES:
To assess the immunogenicity of HBV-002 | 38 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jay Winship, M.D., Study Director — Hawaii Biotech
Locations (1):
- Covance Clinical Research Unit, Honolulu, Hawaii, United States